CLINICAL TRIAL: NCT02049411
Title: Changes of the Short Portable Mental Status Questionnaire (SPMSQ-E) After Ketamine Administration on Ophthalmic Surgery in Geriatric Population.
Brief Title: Ketamine and Changes of the Short Portable Mental Status Questionnaire
Acronym: SPMSQ-E
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: National Polytechnic Institute, Mexico (Other)
Responsible Party: Principal Investigator, Dulce Maria Rascon Martinez, Anesthesiology - Pain Clinical professor., Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R-2012-3601-56
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Ketamine; acute cognitive dysfunction; geriatric patients
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine group (Experimental): Ketamine: (dose 0.3 mcg/kg) included in physiological solution at 0.9% (250 ml) during 2 hours, intravenously.
  Interventions: Drug: Ketamine; Drug: physiological solution
- physiological solution (Sham Comparator): Control group: only physiological solution at 0.9% (250 ml) during 2 hours, intravenously.
  Interventions: Drug: physiological solution

INTERVENTIONS:
Drug: Ketamine — Ketamine: (dose 0.3 mcg/kg) included in physiological solution at 0.9% (250 ml) during 2 hours, intravenously.
  Other Names: Ketalin; Ketalar; Ketanest
  Arms: Ketamine group
Drug: physiological solution — physiological solution at 0.9% (250 ml) during 2 hours, intravenously, with the same physical characteristics of ketamine.
  Other Names: Control; Placebo

SUMMARY:
- Cognitive changes are related to aging, affecting the performance of older patients in the solution of problems and the execution of tasks.

This phenomenon has been observed as a decline of neurophysiological domains, especially memory, and the velocity of thought.

* Anesthesia and surgery performed contributes to its development then, is named post-operative cognitive dysfunction (POCD). The incidence varies due to conditions of:

  1. Anesthesia and surgery.
  2. The time elapsed after surgery.
  3. The population studied, and the type of cognitive test employed.
* The aim of this study is to evaluate the changes around the Short Portable Mental Status Questionnaire (SPMSQ-E) after ketamine administration on ophthalmic surgery on the common conditions of geriatric patients, -comorbid and settings as minor surgery-.

DETAILED DESCRIPTION:
Participants will be patients programmed for a vitrectomy or cataract surgery involving a retrobulbar block, to be carried out with a local anesthesia.

- Administration of ketamine will be suspended during the study for any cause considered as a risk to the patient according to the judgment of the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Patients be over 60 years and older.
* Intraocular pressure less than 20 millimeter of mercury.
* American Society of Anaesthesiologists (ASA) physical status classification, I-III.

Exclusion Criteria:

* History of psychosis or schizophrenia.
* Nephropathy.
* Difficult to control hypertension.
* Uncontrolled hepatic disorders.
* Allergy to ketamine.
* Moderate to severe depression.
* Post-operative delirium.
* Needed to use medications other than those contemplated in the study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to postoperative endpoint error scores on the Short Portable Mental Status Questionnaire (SPMSQ) in both groups | Baseline, 2 hours after surgery
  Patients were included in an analysis of mean change from preoperative to postoperative assessment of the number of items missed on the SPMSQ using analysis of covariance (ANCOVA) model which contained baseline status as covariate, and the treatment group as the effect of interest.

SECONDARY OUTCOMES:
Change in Hemodynamic measures | Baseline, after Retrobulbar block , 90 minutes into surgery.
  Analysis of changes over time in hemodynamic parameters was done during the surgery
Change in respiratory rate measures | Baseline, after Retrobulbar block , 90 minutes into surgery.
  Analysis of changes over time in respiratory rate was done during the surgery with a general lineal model.
Changes in oxygen saturation measures | Baseline, after Retrobulbar block , 90 minutes into surgery.
  Analysis of changes over time in oxygen saturation measures was done during the surgery with a general lineal model
Change in Ramsey Sedation Scale | Baseline, after retrobulbar block, 90 minutes into surgery
  Sedation according to the Ramsey Scale from baseline to the final assessment (90minutes into surgery), was done with a general lineal model.
Change on intraocular pressure measures | Baseline (previous Retrobulbar block), end of surgery.
  Analysis of change in intraocular pressure over time was done previous retrobulbar block and at the end of surgery with a general lineal model over non-surgical eye.
Analgesia | Changes in analgesia after regional anaesthesia (retrobulbar block). Changes in analgesia over 30 minutes after surgery.
  Analgesia was evaluated after regional anesthesia (retrobulbar block) and after surgery, a comparison was made between groups by the Chi-squared test (χ2).

CONTACTS AND LOCATIONS:
Overall Officials: Dulce M. Rascon, M.D, Principal Investigator — Instituto Mexicano del Seguro Social; Maria E. Ocharan, PhD., Study Director — Instituto Politecnico Nacional; Ana Fresan, PhD., Study Chair — Instituto Nacional de Psiquiatria; Jorge H. Genis, Geriatrician, Study Chair — Instituto Mexicano del Seguro Social; Antonio Castellanos, M.D., Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Centro Medico Nacional Siglo XXI. UMAE Hospital de Especialidades, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Tolep K, Higgins N, Muza S, Criner G, Kelsen SG. Comparison of diaphragm strength between healthy adult elderly and young men. Am J Respir Crit Care Med. 1995 Aug;152(2):677-82. doi: 10.1164/ajrccm.152.2.7633725.
- [Background] Phillips-Bute B, Mathew JP, Blumenthal JA, Grocott HP, Laskowitz DT, Jones RH, Mark DB, Newman MF. Association of neurocognitive function and quality of life 1 year after coronary artery bypass graft (CABG) surgery. Psychosom Med. 2006 May-Jun;68(3):369-75. doi: 10.1097/01.psy.0000221272.77984.e2. PMID 16738066
- [Background] Jones MJ, Piggott SE, Vaughan RS, Bayer AJ, Newcombe RG, Twining TC, Pathy J, Rosen M. Cognitive and functional competence after anaesthesia in patients aged over 60: controlled trial of general and regional anaesthesia for elective hip or knee replacement. BMJ. 1990 Jun 30;300(6741):1683-7. doi: 10.1136/bmj.300.6741.1683. PMID 2390547
- [Background] Tsai TL, Sands LP, Leung JM. An Update on Postoperative Cognitive Dysfunction. Adv Anesth. 2010;28(1):269-284. doi: 10.1016/j.aan.2010.09.003. No abstract available. PMID 21151735
- [Background] Caba F, Echevarria M, Cruz A, Rodriguez E, Llamas JM, Martinez MD, Rodriguez R. [Postoperative mental confusion in the elderly with hip fracture. Perioperative risk factors]. Rev Esp Anestesiol Reanim. 1994 Sep-Oct;41(5):255-61. Spanish. PMID 7991903
- [Background] Malouf R, Areosa Sastre A. Vitamin B12 for cognition. Cochrane Database Syst Rev. 2003;(3):CD004326. doi: 10.1002/14651858.CD004326. PMID 12918012
- [Background] Balk EM, Raman G, Tatsioni A, Chung M, Lau J, Rosenberg IH. Vitamin B6, B12, and folic acid supplementation and cognitive function: a systematic review of randomized trials. Arch Intern Med. 2007 Jan 8;167(1):21-30. doi: 10.1001/archinte.167.1.21. PMID 17210874
- [Background] Hudetz JA, Pagel PS. Neuroprotection by ketamine: a review of the experimental and clinical evidence. J Cardiothorac Vasc Anesth. 2010 Feb;24(1):131-42. doi: 10.1053/j.jvca.2009.05.008. Epub 2009 Jul 29. No abstract available. PMID 19640746
- [Background] Faden AI, Demediuk P, Panter SS, Vink R. The role of excitatory amino acids and NMDA receptors in traumatic brain injury. Science. 1989 May 19;244(4906):798-800. doi: 10.1126/science.2567056.
- [Background] Hartvig P, Valtysson J, Lindner KJ, Kristensen J, Karlsten R, Gustafsson LL, Persson J, Svensson JO, Oye I, Antoni G, et al. Central nervous system effects of subdissociative doses of (S)-ketamine are related to plasma and brain concentrations measured with positron emission tomography in healthy volunteers. Clin Pharmacol Ther. 1995 Aug;58(2):165-73. doi: 10.1016/0009-9236(95)90194-9. PMID 7648766
- [Background] Pfeiffer E. A short portable mental status questionnaire for the assessment of organic brain deficit in elderly patients. J Am Geriatr Soc. 1975 Oct;23(10):433-41. doi: 10.1111/j.1532-5415.1975.tb00927.x. PMID 1159263
- [Background] Gonzalez Montalvo J I; Rodriguez L; Ruiperez I. Validacion del cuestionario de Pfeiffer y la escala de incapacidad mental de la cruz roja en la deteccion del deterioro mental en los pacientes externos de un servicio de Geriatria. Revista Española de Geriatría y Gerontología. 1991, 27 (3): 129-133.
- [Background] Attix Deborah K, Welsh-Bohmer Kathleen A: Geriatric Neuropsychology: assessment and intervention. Guilford Press, 2006.
- [Result] Hudetz JA, Iqbal Z, Gandhi SD, Patterson KM, Byrne AJ, Hudetz AG, Pagel PS, Warltier DC. Ketamine attenuates post-operative cognitive dysfunction after cardiac surgery. Acta Anaesthesiol Scand. 2009 Aug;53(7):864-72. doi: 10.1111/j.1399-6576.2009.01978.x. Epub 2009 Apr 28. PMID 19422355
- [Result] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Result] Malhotra AK, Pinals DA, Weingartner H, Sirocco K, Missar CD, Pickar D, Breier A. NMDA receptor function and human cognition: the effects of ketamine in healthy volunteers. Neuropsychopharmacology. 1996 May;14(5):301-7. doi: 10.1016/0893-133X(95)00137-3. PMID 8703299
- [Result] Krystal JH, Karper LP, Seibyl JP, Freeman GK, Delaney R, Bremner JD, Heninger GR, Bowers MB Jr, Charney DS. Subanesthetic effects of the noncompetitive NMDA antagonist, ketamine, in humans. Psychotomimetic, perceptual, cognitive, and neuroendocrine responses. Arch Gen Psychiatry. 1994 Mar;51(3):199-214. doi: 10.1001/archpsyc.1994.03950030035004. PMID 8122957
- [Result] Roytblat L, Talmor D, Rachinsky M, Greemberg L, Pekar A, Appelbaum A, Gurman GM, Shapira Y, Duvdenani A. Ketamine attenuates the interleukin-6 response after cardiopulmonary bypass. Anesth Analg. 1998 Aug;87(2):266-71. doi: 10.1097/00000539-199808000-00006. PMID 9706914
- [Result] Bartoc C, Frumento RJ, Jalbout M, Bennett-Guerrero E, Du E, Nishanian E. A randomized, double-blind, placebo-controlled study assessing the anti-inflammatory effects of ketamine in cardiac surgical patients. J Cardiothorac Vasc Anesth. 2006 Apr;20(2):217-22. doi: 10.1053/j.jvca.2005.12.005. Epub 2006 Mar 9. PMID 16616662 (Retraction: PMID 25319992 J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1435)
- [Result] Vollenweider FX, Leenders KL, Oye I, Hell D, Angst J. Differential psychopathology and patterns of cerebral glucose utilisation produced by (S)- and (R)-ketamine in healthy volunteers using positron emission tomography (PET). Eur Neuropsychopharmacol. 1997 Feb;7(1):25-38. doi: 10.1016/s0924-977x(96)00042-9. PMID 9088882
- [Result] Holcomb HH, Lahti AC, Medoff DR, Weiler M, Tamminga CA. Sequential regional cerebral blood flow brain scans using PET with H2(15)O demonstrate ketamine actions in CNS dynamically. Neuropsychopharmacology. 2001 Aug;25(2):165-72. doi: 10.1016/S0893-133X(01)00229-9. PMID 11425500
- [Result] Lahti AC, Koffel B, LaPorte D, Tamminga CA. Subanesthetic doses of ketamine stimulate psychosis in schizophrenia. Neuropsychopharmacology. 1995 Aug;13(1):9-19. doi: 10.1016/0893-133X(94)00131-I. PMID 8526975
- [Result] Takeshita H, Okuda Y, Sari A. The effects of ketamine on cerebral circulation and metabolism in man. Anesthesiology. 1972 Jan;36(1):69-75. doi: 10.1097/00000542-197201000-00013. No abstract available. PMID 5006989
- [Result] O'Neill LA, Kaltschmidt C. NF-kappa B: a crucial transcription factor for glial and neuronal cell function. Trends Neurosci. 1997 Jun;20(6):252-8. doi: 10.1016/s0166-2236(96)01035-1. PMID 9185306
- [Result] Shen C, Nettleton D, Jiang M, Kim SK, Powell-Coffman JA. Roles of the HIF-1 hypoxia-inducible factor during hypoxia response in Caenorhabditis elegans. J Biol Chem. 2005 May 27;280(21):20580-8. doi: 10.1074/jbc.M501894200. Epub 2005 Mar 21. PMID 15781453
- [Result] Sakai T, Ichiyama T, Whitten CW, Giesecke AH, Lipton JM. Ketamine suppresses endotoxin-induced NF-kappaB expression. Can J Anaesth. 2000 Oct;47(10):1019-24. doi: 10.1007/BF03024876. PMID 11032280
- [Result] Baldwin AS Jr. The NF-kappa B and I kappa B proteins: new discoveries and insights. Annu Rev Immunol. 1996;14:649-83. doi: 10.1146/annurev.immunol.14.1.649. PMID 8717528
- [Result] Kochs E, Werner C, Hoffman WE, Mollenberg O, Schulte am Esch J. Concurrent increases in brain electrical activity and intracranial blood flow velocity during low-dose ketamine anaesthesia. Can J Anaesth. 1991 Oct;38(7):826-30. doi: 10.1007/BF03036955. PMID 1742815
- [Result] Langsjo JW, Kaisti KK, Aalto S, Hinkka S, Aantaa R, Oikonen V, Sipila H, Kurki T, Silvanto M, Scheinin H. Effects of subanesthetic doses of ketamine on regional cerebral blood flow, oxygen consumption, and blood volume in humans. Anesthesiology. 2003 Sep;99(3):614-23. doi: 10.1097/00000542-200309000-00016. PMID 12960545
- [Result] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Result] Kudoh A, Takahira Y, Katagai H, Takazawa T. Small-dose ketamine improves the postoperative state of depressed patients. Anesth Analg. 2002 Jul;95(1):114-8, table of contents. doi: 10.1097/00000539-200207000-00020. PMID 12088953
- [Result] Sadove MS, Shulman M, Hatano S, Fevold N. Analgesic effects of ketamine administered in subdissociative doses. Anesth Analg. 1971 May-Jun;50(3):452-7. No abstract available. PMID 5103784
- [Result] Bell RF. Ketamine for chronic non-cancer pain. Pain. 2009 Feb;141(3):210-214. doi: 10.1016/j.pain.2008.12.003. Epub 2009 Jan 6. No abstract available. PMID 19128879
- [Result] Vlaeyen JWS, Linton SJ. Are we "fear-avoidant"? Pain. 2006 Oct;124(3):240-241. doi: 10.1016/j.pain.2006.06.031. Epub 2006 Aug 9. No abstract available. PMID 16901646
- [Result] Loots H, Wiseman R. Ophthalmic anaesthesia, agents for sedation in ophthalmic surgery: A review of the pharmacodynamics and clinical applications. Current Anaesthesia& Critical Care (2006) 17, 179-190
- [Result] Frey K, Sukhani R, Pawlowski J, Pappas AL, Mikat-Stevens M, Slogoff S. Propofol versus propofol-ketamine sedation for retrobulbar nerve block: comparison of sedation quality, intraocular pressure changes, and recovery profiles. Anesth Analg. 1999 Aug;89(2):317-21. doi: 10.1097/00000539-199908000-00013. PMID 10439740
- [Result] Santiveri X, Molto L, Rodriguez C, Sandin F, Vilaplana J, Castillo J. [Sedation and analgesia with propofol plus low-dose ketamine for retrobulbar block]. Rev Esp Anestesiol Reanim. 2006 Nov;53(9):545-9. Spanish. PMID 17297830
- [Result] Moorthy SS, Valluri S, Cummings L. Retrobulbar anesthesia. Ophthalmology. 2002 Jan;109(1):5-6. doi: 10.1016/s0161-6420(01)00911-3. No abstract available. PMID 11772567
- [Result] Slogoff S, Allen GW, Wessels JV, Cheney DH. Clinical experience with subanesthetic ketamine. Anesth Analg. 1974 May-Jun;53(3):354-8. No abstract available. PMID 4856927